CLINICAL TRIAL: NCT05935657
Title: The Effect of Remimazolam and Dexmedetomidine on the Incidence of Hypotension During Spinal Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Gyeong-Jo Byeon, MD, PhD, Associate professor for fund, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20230608
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Remimazolam; Spinal Anesthesia
MeSH Terms: interventions — remimazolam; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Group (Experimental): sedation with remimazolam
  Interventions: Drug: Remimazolam
- Dexmedetomidine group (Active Comparator): sedation with dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Remimazolam — 0.075 mg/kg Remimazolam bolus infusion for 1 min, then 0.1~1.0 mg/kg/h continuous infusion
  Other Names: Byfavo
  Arms: Remimazolam Group
Drug: Dexmedetomidine — 1 mcg/kg Dexmedetomidine infusion for 10 min, then 0.2~0.7 mcg/kg/h continuous infusion
  Other Names: Precedex
  Arms: Dexmedetomidine group

SUMMARY:
The goal of this clinical trial is to compare the effect of remimazolam and dexmedetomidine on the incidence of hypotension during spinal anesthesia in adult patients.

DETAILED DESCRIPTION:
Sedation during spinal anesthesia can reduce the patient's anxiety and increase satisfaction, but sedatives such as dexmedetomidine and midazolam may cause hemodynamic instability such as hypotension and bradycardia. In previous studies , hypotension occurred in about 33% and bradycardia in about 13% during spinal anesthesia, which is related to reduced cardiac output due to sympathetic blockade and relative activation of the parasympathetic nerve.

In the study comparing remimazolam and dexmedetomidine in patients with delirium after orthopedic surgery, the incidence of hypotension was lower in the remimazolam group (10.8%) than in the dexmedetomidine group (39.5%) (p=0.007) and there was no significant difference between the remimazolam group (2.7%) and the dexmedetomidine group (13.2%) in the incidence of bradycardia (p=0.200).

However, the effect of remimazolam on the incidence of hypotension during spinal anesthesia has not been revealed. Therefore, this study is designed to compare the effect of remimazolam and dexmedetomidine on the incidence of hypotension during spinal anesthesia in adults patients.

ELIGIBILITY:
Inclusion Criteria:

- Patient scheduled for surgery under spinal anesthesia, aged 19-79, of ASA class I, II, or III

Exclusion Criteria:

* Patient refusal
* Contraindications to regional or neuraxial anesthesia (patient refusal, increased intracranial pressure, infection at puncture site, underlying neurologic disease, severe hypovolemia, severe aortic or mitral stenosis, thrombocytopenia or coagulopathy, sepsis)
* Contraindications or allergy to dexmedetomidine or remimazolam administration
* Emergency surgery
* Pregnancy

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of intraoperative hypotension | Intraoperative period
  mean blood pressure lower than 65 mmHg or systolic blood pressure lower than 80% of baseline

SECONDARY OUTCOMES:
Incidence of intraoperative bradycardia | Intraoperative period
  heart rate lower than 45 bpm
Incidence of intraoperative hypertension | Intraoperative period
  mean blood pressure higher than 120 mmHg or systolic blood pressure higher than 120% of baseline
Incidence of respiratory depression | Intraoperative period
  respiratory rate lower than 8 per minute
Incidence of hypoxia | Intraoperative period
  oxygen saturation detected by pulse oxymetry less than 93%
Intraoperative Ramsay sedation scale | Intraoperative period
  score of 1~6
Number of phenylephrine, ephedrine, atropine administered | Intraoperative period
  number of administration

CONTACTS AND LOCATIONS:
Overall Officials: Gyengjo Byeon, PhD, Study Director — Pusan National University Yangsan Hospital